CLINICAL TRIAL: NCT05240053
Title: Enhanced Recovery Program After Laparoscopic Colorectal Surgery During The Era Of COVID-19 : A Randomized Controlled Trial
Brief Title: Enhanced Recovery Program After Laparoscopic Colorectal Surgery During The Era Of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: zagazig general surgey departe
Record Dates: First submitted 2022-02-11; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Disorders
Keywords: enhanced oral recovery; , colorectal disorders

STUDY DESIGN:
Intervention Model Description: The investigators included all patients who were subjected to laparoscopic colorectal surgery at our center between ( December 2019 to December 2021) for benign & malignant conditions. sample size was 50 patients , divided into 2 equal groups . Group 1: included 25 patients who were subjected to enhance recovery program after laparoscopic colorectal surgery . Group 2: included 25 patients who were subjected to traditional way - nothing by mouth until the resolution of ileus, then a fluid diet, followed by a regular diet after laparoscopic colorectal surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Active Comparator): Group 1: included 25 patients who were subjected to enhance recovery program after laparoscopic colorectal surgery .
  Interventions: Other: enhanced recovery programe
- group (2) (No Intervention): Group 2: included 25 patients who were subjected to traditional way

INTERVENTIONS:
Other: enhanced recovery programe — Early postoperative analgesia , early oral intake , early mobilization , early removal of nasogastric tube & drains if any. The patients in this group started clear fluid once they awaked from anesthesia , a full liquid diet on first postoperative day , normal diet on second day provided that there was no vomiting or abdominal distension. The patients in this group were instructed for early ambulation & encouraged to stay out of the bed for 4 hours on first day postoperative , 6 hours in following day , 8 hours on subsequent days. Also they were encouraged to walk the length of 3 meters once on first day postoperative , twice on day 2 & three times on subsequent days. Regarding analgesia in this group postoperatively , they were received fentanyl via an epidural catheter.
  Arms: group (1)

SUMMARY:
The investigators included all patients who were subjected to laparoscopic colorectal surgery at investigators' center between ( December 2019 to December 2021) for benign & malignant conditions. sample size was 50 patients , divided into 2 equal groups . Group 1: included 25 patients who were subjected to enhance recovery program after laparoscopic colorectal surgery . Group 2: included 25 patients who were subjected to traditional way - nothing by mouth until the resolution of ileus, then a fluid diet, followed by a regular diet after laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
The investigators included all patients who were subjected to laparoscopic colorectal surgery at investigators' center between ( December 2019 to December 2021) for benign & malignant conditions. The study was approved by the research and Ethics committee of our university and performed in accordance with the code of ethics of the world medical association (Declaration of Helsinki) for studies involving humans. A written informed consent was obtained from all participants.

Sample size The sample size was calculated using open Epi program . sample size was 50 patients , divided into 2 equal groups . Group 1: included 25 patients who were subjected to enhance recovery program after laparoscopic colorectal surgery . Group 2: included 25 patients who were subjected to traditional way - nothing by mouth until the resolution of ileus, then a fluid diet, followed by a regular diet after laparoscopic colorectal surgery.

Perioperative measures:

In this prospective randomized controlled trials , all patients were subjected to the followings: patients were selected by randomization method , Full history taking , Complete physical examination , laboratory investigations ( complete blood picture , liver and kidney functions , coagulation profile , tumor marker tests, serum electrolytes) , patients were assessed radio- logically by barium enema, abdominal ultrasound ,pelvic and abdominal CT, bone survey and chest X-ray in addition to colonoscopy and biopsy for diagnosis of colorectal cancer, all cases were well prepared by correction of electrolytes and acid-base disturbance , all cases were subjected to colonic preparation.

Surgical techniques :

Group (1) : 25 patients were subjected to enhanced recovery program after laparoscopic colorectal surgery for either benign or malignant condition including different types of anastomosis either handmade or staplers assisted. They were informed about the program and what was to happen during hospitalization , food intake , ambulation after surgery , fasting 2 hours for liquid & 6 hours for solid. Prophylactic antibiotic was given . also thromboembolism prophylaxis was given . Good nutrition for the patients was achieved .both crystalloid & colloid with vasopressor were given intraoperative with caution to keep intraoperative fluid less than 3000-3500ml with no use of drains & nasogastric tube if possible or as can as possible. Early postoperative analgesia , early oral intake , early mobilization , early removal of nasogastric tube & drains if any. The patients in this group started clear fluid once they awaked from anesthesia , a full liquid diet on first postoperative day , normal diet on second day provided that there was no vomiting or abdominal distension. The patients in this group were instructed for early ambulation & encouraged to stay out of the bed for 4 hours on first day postoperative , 6 hours in following day , 8 hours on subsequent days. Also they were encouraged to walk the length of 3 meters once on first day postoperative , twice on day 2 & three times on subsequent days. Regarding analgesia in this group postoperatively , they were received fentanyl via an epidural catheter.

Group (2) : included 25 patients who were subjected to conventional rehabilitation program after laparoscopic colorectal resection for benign or malignant conditions . they were subjected to nothing per mouth for 5 days until resolution of ileus , fluid diet followed by usual diet . patients were mobilized by nurses according to patient wellness . instructions about importance of mobilization were given to the patients. Pain was managed in this group by paracetamol & non- steroidal anti-inflammatory drug (NSAID) infusion .

Patients in both groups were eligible for discharge when they were self-caring, were tolerating oral fluid and diet, had bowel function, and were independently mobile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ranged from 20-75 years
* patients who had no contraindication for laparoscopic surgery
* good general condition with American society of anesthesiology (ASA) I & II

Exclusion Criteria:

* patients who had bad general condition (ASA ≥3)
* patients with age above 75 years
* patients with uncompensated cardiopulmonary disease , immunological disorders ,immunosuppressive therapy for any cause.
* Patients who had chronic liver disease
* patients who underwent emergency laparotomy and had a stoma created for them or those with metastasis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
incidence of complications after enhanced recovery program | within one week after the surgery
  incidence of complications after after enhanced recovery program

SECONDARY OUTCOMES:
incidence of mortality after enhanced recovery program | within one month after the surgery
  incidence of mortality after enhanced recovery program

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — ZAGAZIG UNIVERSITY HOSPITALS
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqua, Egypt